CLINICAL TRIAL: NCT03211247
Title: A Double-blind, Placebo-controlled, Randomized Phase III Trial to Assess the Safety and Efficacy of Viaskin Peanut in Peanut-allergic Young Children 1-3 Years of Age.
Brief Title: Safety and Efficacy Study of Viaskin Peanut in Peanut-allergic Young Children 1-3 Years of Age
Acronym: EPITOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPITOPE
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Peanut Allergy
Keywords: EPIT; Epicutaneous; Immunotherapy; Viaskin
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A Viaskin Peanut 250 mcg (Experimental)
  Interventions: Biological: Part A Viaskin Peanut 250 mcg
- Part A Viaskin Peanut 100 mcg (Experimental)
  Interventions: Biological: Part A Viaskin Peanut 100 mcg
- Part A Placebo (Placebo Comparator)
  Interventions: Biological: Part A Placebo
- Part B Viaskin Peanut 250 mcg (Experimental)
  Interventions: Biological: Part B Viaskin Peanut 250 mcg
- Part B Placebo (Placebo Comparator)
  Interventions: Biological: Part B Placebo

INTERVENTIONS:
Biological: Part A Viaskin Peanut 250 mcg — Viaskin Peanut 250 mcg, once daily
  Arms: Part A Viaskin Peanut 250 mcg
Biological: Part A Viaskin Peanut 100 mcg — Viaskin Peanut 100 mcg, once daily
  Arms: Part A Viaskin Peanut 100 mcg
Biological: Part A Placebo — Placebo patch, once daily
  Arms: Part A Placebo
Biological: Part B Viaskin Peanut 250 mcg — Viaskin Peanut 250 mcg, once daily
  Arms: Part B Viaskin Peanut 250 mcg
Biological: Part B Placebo — Placebo patch, once daily
  Arms: Part B Placebo

SUMMARY:
The study aims to assess the safety and efficacy of Viaskin Peanut to induce desensitization to peanut in peanut-allergic children 1 to 3 years of age after a 12-month treatment by EPicutaneous ImmunoTherapy (EPIT).

DETAILED DESCRIPTION:
The study comprised of two parts:

* In part A, subjects were randomized to receive either Viaskin Peanut 250 mcg, or Viaskin Peanut 100 mcg or the placebo in a 2:1 ratio, for 12 months. After 3 months of treatment, a data safety monitoring board had to determine the active dose to be applyed during the part B
* In Part B, subjects were randomized to receive either Viaskin Peanut 250 mcg or the placebo in a 2:1 ratio, for 12 months

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female from 1-3 years of age;
* Physician-diagnosed peanut allergy;
* Peanut-specific IgE level > 0.7 kU/L;
* Positive peanut SPT with a largest wheal diameter ≥ 6 mm;
* Positive DBPCFC at ≤ 300 mg peanut protein;

Key Exclusion Criteria:

* Uncontrolled asthma;
* History of severe anaphylaxis to peanut;
* Prior immunotherapy to any food or other immunotherapy;
* Generalized severe dermatologic disease;

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 414 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (27):
  - University of Arizona Health Science, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California School of Medicine, Los Angeles, California
  - University of California, Rady Children's Hospital, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's national Health System, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of CHicago, Chicago, Illinois
  - The Universal of Chicago Medical Center, Chicago, Illinois
  - Riley Hospital for Children at Indiana University, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Childrens' Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - The University of North Carolina - Chapell Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - ASTHMA, Inc., Seattle, Washington
- Australia (6):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Sydney Children's Hospital, Randwick, NWS
  - Queensland Children's Hospital, South Brisbane, Queensland
  - The Women's and children's hospital, North Adelaide, South Australia
  - The Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
  - CHUM & CHU Sainte-Justine, Montreal, Quebec
- France (5):
  - CHRU Lille, Lille
  - CHRU Metz-Thionville, Metz
  - Hopitaux Pediatriques de Nice, Nice
  - Hopital Necker, Paris
  - CHRU Nancy, Vandœuvre-lès-Nancy
- Germany (3):
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitatklinikum Giessen und Marburg, Marburg
- Cork University Hospital, Cork, Ireland
- Erasmus MC Sophia Children's Hospital, Rotterdam, Netherlands
- United Kingdom (5):
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - St.Mary's Hospital, London
  - ROyal Manchester Children's Hospital, Manchester
  - Sheffield Children's Hospital, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scurlock AM, Fleischer DM, Toit GD, Arends NJT, Pongracic JA, Trujillo J, Turner P, Vogelberg C, Bee KJ, Green TD, Meney J, Bois T, Campbell DE, Sampson HA, Burks AW. Efficacy and safety of epicutaneous immunotherapy in children with peanut allergy with atopic comorbidities. Ann Allergy Asthma Immunol. 2025 Aug;135(2):203-210. doi: 10.1016/j.anai.2025.04.002. Epub 2025 Apr 7. PMID 40204253
- [Derived] Greenhawt M, Sindher SB, Wang J, O'Sullivan M, du Toit G, Kim EH, Albright D, Anvari S, Arends N, Arkwright PD, Begin P, Blumchen K, Bourrier T, Brown-Whitehorn T, Cassell H, Chan ES, Ciaccio CE, Deschildre A, Divaret-Chauveau A, Dorris SL, Dorsey MJ, Eiwegger T, Erlewyn-Lajeunesse M, Fleischer DM, Ford LS, Garcia-Lloret M, Giovannini-Chami L, Hourihane JO, Jay N, Jones SM, Kerns LA, Kloepfer KM, Leonard S, Lezmi G, Lieberman JA, Lomas J, Makhija M, Parrish C, Peake J, Perrett KP, Petroni D, Pfutzner W, Pongracic JA, Quinn P, Robison RG, Sanders G, Schneider L, Sharma HP, Trujillo J, Turner PJ, Tuttle K, Upton JE, Varshney P, Vickery BP, Vogelberg C, Wainstein B, Wood RA, Bee KJ, Campbell DE, Green TD, Rouissi R, Peillon A, Bahnson HT, Bois T, Sampson HA, Burks AW. Phase 3 Trial of Epicutaneous Immunotherapy in Toddlers with Peanut Allergy. N Engl J Med. 2023 May 11;388(19):1755-1766. doi: 10.1056/NEJMoa2212895. PMID 37163622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III was conducted in participants aged 1 to 3 years with peanut-allergy at 51 centers in Australia, Canada, Europe, and the United States of America. The entire duration of study was approximately 62 weeks (6-week: screening period; 12-month treatment period; and 4-week follow-up period).
Pre-assignment Details: In Part A, a total of 51 participants were randomized either in the placebo arm or in the 2 active arms (Viaskin Peanut (DBV712) 100 mcg or 250 mcg) in a 1:2:2 ratio.
  In Part B, a total of 362 participants were randomized in a 2:1 ratio to receive Viaskin Peanut (DBV712) 250 mcg or placebo.
Groups:
- Part B Viaskin Peanut 250 mcg; Part A Viaskin Peanut 250 mcg: Participants applied 1 new Viaskin Peanut 250 mcg patch on intact skin for 24 hours daily for up to 12 months. Each patch contained 250 mcg peanut protein extract for epicutaneous administration. The application duration was progressively increased to a duration of 24 ±4 hours daily over a 4-week period (2 hours during the first week, 4 hours during the second week, 8 hours during the third week, 12 hours during the fourth week onwards, and 24 ± 4 hours every day fifth week onwards).
- Part B Placebo; Part A Placebo: Participants applied 1 new placebo patch on intact skin for 24 hours daily for up to 12 months. The application duration was progressively increased to a duration of 24 ±4 hours daily over a 4-week period (2 hours during the first week, 4 hours during the second week, 8 hours during the third week, 12 hours during the fourth week onwards, and 24 ± 4 hours every day fifth week onwards).
- Part A Viaskin Peanut 100 mcg: Participants applied 1 new Viaskin Peanut 100 mcg patch on intact skin for 24 hours daily for up to 12 months. Each patch contained 100 mcg peanut protein extract for epicutaneous administration. The application duration was progressively increased to a duration of 24 ±4 hours daily over a 4-week period (2 hours during the first week, 4 hours during the second week, 8 hours during the third week, 12 hours during the fourth week onwards, and 24 ± 4 hours every day fifth week onwards).
Period: Overall Study
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
Started | 244 | 118 | 21 | 20 | 10
Completed | 208 | 99 | 17 | 16 | 9
Not Completed | 36 | 19 | 4 | 4 | 1
Not completed — Adverse Event | 8 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 2 | 0 | 0 | 0 | 0
Not completed — Participant withdrawal by Parent or Caregiver | 18 | 13 | 2 | 1 | 0
Not completed — Participant did not want to complete oral food challenge | 5 | 2 | 1 | 3 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised of all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo | Total
Number analyzed (Participants) | 244 | 118 | 21 | 20 | 10 | 413
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 244 | 118 | 21 | 20 | 10 | 413
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 34 | 8 | 5 | 4 | 130
  Male | 165 | 84 | 13 | 15 | 6 | 283
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 159 | 70 | 15 | 17 | 7 | 268
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2
  Asian | 41 | 24 | 1 | 2 | 1 | 69
  Other | 35 | 17 | 5 | 1 | 2 | 60
  Not collected | 8 | 6 | 0 | 0 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Responders at Month 12
Description: A participant was defined as a treatment responder if the initial eliciting dose (ED) was > 10 milligram (mg) peanut protein and the ED was ≥1000 mg peanut protein at the post-treatment double-blind placebo-controlled food challenge (DBPCFC) at Month 12 OR the initial ED at baseline was ≤10 mg peanut protein and the ED was ≥300 mg peanut protein at the post-treatment DBPCFC at Month 12.
Time Frame: Month 12
Population: The FAS comprised of all participants who were randomized in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
Number analyzed (Participants) | 244 | 118 | 21 | 20 | 10
Percentage of participants | 67.0 [60.93 to 73.01] | 33.5 [24.84 to 42.24] | 52.4 [29.8 to 74.3] | 70.0 [45.7 to 88.1] | 60.0 [26.2 to 74.3]
Statistical Analysis 1: Comparison: Part B Viaskin Peanut 250 mcg vs Part B Placebo; Analysis of the difference in response rates between DBV712 250 μg group and Placebo group and 2-sided Farrington-Manning 95% confidence interval (CI). P-value was obtained from a 2-sided 5% test to evaluate the null hypothesis of no difference in response rates between treatment groups using the Wald method. Clinical relevance was evaluated based on the lower bound of the Farrignton-Manning 95% CI of the difference in response rates ≥15%; Test type: Other; p < 0.001, Wald test; Proportion difference = 33.4, 95% CI 2-sided [22.36 to 44.49] — The 2-sided Farrington-Manning 95% confidence interval for the difference in response rates was calculated

2. Secondary Outcome: Cumulative Reactive Dose (CRD) of Peanut Protein at Month 12 Using Analysis of Covariance (ANCOVA) Model
Description: The peanut protein CRD was defined as the sum of all peanut protein doses taken by the participant during the DBPCFC, calculated as follows:
  If the ED reported by the investigator in the electronic case report form (eCRF) is missing, then the CRD is missing; If the ED reported by the investigator in the eCRF was not missing then the CRD was calculated as the sum of all doses given, including also the partial doses. The CRD in each treatment group at Month 12 was compared using ANCOVA model.
Time Frame: Month 12
Population: The FAS comprised of all participants who were randomized in the study.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: milligram (mg)
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
Number analyzed (Participants) | 244 | 118 | 21 | 20 | 10
milligram (mg) | 1010.31 [842.18 to 1212.01] | 322.57 [248.37 to 418.94] | 788.74 [220.20 to 2825.24] | 1155.90 [367.53 to 3635.38] | 1153.47 [474.34 to 2804.91]

3. Secondary Outcome: Change From Baseline in CRD of Peanut Protein to Month 12
Description: The peanut protein CRD was defined as the sum of all peanut protein doses taken by the participant during the DBPCFC, calculated as follows:
  If the ED reported by the investigator in the eCRF is missing, then the CRD is missing; If the ED reported by the investigator in the eCRF was not missing then the CRD was calculated as the sum of all doses given, including also the partial doses.
Time Frame: Baseline (Day 1) and Month 12
Population: The FAS comprised of all participants who were randomized in the study.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
Number analyzed (Participants) | 244 | 118 | 21 | 20 | 10
mg | 1300.0 [140.0 to 3000.0] | 0.0 [0.0 to 1000.0] | 540.0 [0.0 to 2930.0] | 1250.0 [2.5 to 3000.0] | 1000.0 [300.0 to 2560.0]

4. Secondary Outcome: ED of Peanut Protein at Month 12 Using ANCOVA Model
Description: The peanut protein ED was the individual dose of peanut protein administered to participants during the food challenge procedure, which triggered objective allergic reactions, leading to stopping the challenge. The ED in each treatment group at Month 12 was compared using ANCOVA model.
Time Frame: Month 12
Population: The FAS comprised of all participants who were randomized in the study.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
Number analyzed (Participants) | 244 | 118 | 21 | 20 | 10
mg | 659.36 [553.84 to 784.99] | 223.12 [173.40 to 287.09] | 526.31 [151.15 to 1832.58] | 730.38 [254.17 to 2098.83] | 760.60 [325.34 to 1778.17]

5. Secondary Outcome: Change From Baseline in ED of Peanut Protein to Month 12
Description: The peanut protein ED was the individual dose of peanut protein administered to participants during the food challenge procedure, which triggered objective allergic reactions, leading to stopping the challenge.
Time Frame: Baseline (Day 1) and Month 12
Population: The FAS comprised of all participants who were randomized in the study.
Measure: Median (Inter-Quartile Range); unit: mg
Groups:
- Part A Viaskin Peanut 100 mcg: Participants applied 1 new Viaskin Peanut 250 mcg patch on intact skin for 24 hours daily for up to 12 months. Each patch contained 250 mcg peanut protein extract for epicutaneous administration. The application duration was progressively increased to a duration of 24 ±4 hours daily over a 4-week period (2 hours during the first week, 4 hours during the second week, 8 hours during the third week, 12 hours during the fourth week onwards, and 24 ± 4 hours every day fifth week onwards).
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
Number analyzed (Participants) | 244 | 118 | 21 | 21 | 10
mg | 900.0 [90.0 to 1700.0] | 0.0 [0.0 to 700.0] | 700.0 [0.0 to 1700.0] | 700.0 [0.0 to 1700.0] | 700.0 [200.0 to 1700.0]

6. Secondary Outcome: Percentage of Participants With Severity of Objective Symptoms at Baseline and Month 12 During Double-Blind Placebo-Controlled Food Challenge
Description: The objective symptoms collected during the DBPCFC included skin (erythematous rash, pruritus, urticaria/angioedema, rash), upper respiratory (sneezing/itching, nasal congestion, rhinorrhea, laryngeal), lower respiratory (wheezing), gastrointestinal (diarrhea, vomiting, cardiovascular), and eyes (conjunctivitis, any other objective symptoms), with the exception of erythematous rash (recorded as Yes/No), each symptom was graded as: 0=" absent",1=" mild", 2=" moderate" or 3=" severe". For erythematous rash, the percent area involved was collected. Percentages were calculated based on the number of participants in each time point. Subjective abdominal pain (when graded 2 or 3) was also considered for this analysis.
Time Frame: Baseline (Day 1) and Month 12
Population: The FAS comprised of all participants who were randomized in the study. This outcome was measured on Part B subjects only. Therefore subjects from Part A are reported as zero in the outcome measure data table.
Measure: Number; unit: Percentage of participants
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
Number analyzed (Participants) | 244 | 118 | 0 | 0 | 0
Percentage of participants
  Baseline: Absent | 0 | 0 |  |  |
  Baseline: Mild | 7.0 | 7.6 |  |  |
  Baseline: Moderate | 68.4 | 67.8 |  |  |
  Baseline: Severe | 24.6 | 24.6 |  |  |
  Month 12: Absent: number analyzed (Participants) | 200 | 98 | 0 | 0 | 0
  Month 12: Absent | 16.0 | 6.1 |  |  |
  Month 12: Mild: number analyzed (Participants) | 200 | 98 | 0 | 0 | 0
  Month 12: Mild | 20.5 | 14.3 |  |  |
  Month 12: Moderate: number analyzed (Participants) | 200 | 98 | 0 | 0 | 0
  Month 12: Moderate | 51.0 | 51.0 |  |  |
  Month 12: Severe: number analyzed (Participants) | 200 | 98 | 0 | 0 | 0
  Month 12: Severe | 12.5 | 28.6 |  |  |

ADVERSE EVENTS:
Time Frame: The TEAEs were collected from Day 1 up to Month 12
Description: The SAF comprised of all participants from the FAS who received at least 1 dose of IMP.
Arm/Group | Part B Viaskin Peanut 250 mcg | Part B Placebo | Part A Viaskin Peanut 250 mcg | Part A Viaskin Peanut 100 mcg | Part A Placebo
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/118 | 0/21 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 21/244 | 3/118 | 0/21 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 244/244 | 117/118 | 21/21 | 20/20 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part B Viaskin Peanut 250 mcg (N=244) | Part B Placebo (N=118) | Part A Viaskin Peanut 250 mcg (N=21) | Part A Viaskin Peanut 100 mcg (N=20) | Part A Placebo (N=10)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic Reaction To Food (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medication Error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aplasia Pure Red Cell (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital Edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part B Viaskin Peanut 250 mcg (N=244) | Part B Placebo (N=118) | Part A Viaskin Peanut 250 mcg (N=21) | Part A Viaskin Peanut 100 mcg (N=20) | Part A Placebo (N=10)
Application Site Erythema (General disorders) | 239 (2182) | 107 (760) | 18 (21) | 14 (15) | 6 (13)
Application Site Pruritus (General disorders) | 231 (2925) | 72 (523) | 13 (15) | 11 (29) | 1 (2)
Application Site Swelling (General disorders) | 177 (2044) | 46 (278) | 7 (15) | 2 (3) | 2 (2)
Pyrexia (General disorders) | 84 (150) | 50 (83) | 5 (8) | 6 (11) | 2 (7)
Application Site Oedema (General disorders) | 58 (504) | 21 (105) | 0 (0) | 1 (1) | 0 (0)
Application Site Urticaria (General disorders) | 68 (152) | 3 (3) | 2 (8) | 3 (10) | 0 (0)
Application Site Vesicles (General disorders) | 43 (179) | 11 (21) | 1 (1) | 0 (0) | 1 (2)
Application Site Papules (General disorders) | 41 (63) | 9 (10) | 2 (2) | 0 (0) | 0 (0)
Application Site Eczema (General disorders) | 34 (66) | 10 (12) | 1 (1) | 0 (0) | 0 (0)
Application Site Erosion (General disorders) | 32 (44) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Application Site Discoloration (General disorders) | 15 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Allergy (Immune system disorders) | 33 (63) | 13 (20) | 5 (5) | 4 (6) | 0 (0)
Hypersensitivity (Immune system disorders) | 24 (30) | 11 (22) | 5 (8) | 3 (7) | 0 (0)
Seasonal Allergy (Immune system disorders) | 28 (50) | 3 (4) | 2 (5) | 2 (3) | 2 (4)
Anaphylactic Reaction (Immune system disorders) | 19 (25) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 56 (87) | 21 (34) | 7 (10) | 4 (8) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 22 (48) | 11 (21) | 0 (0) | 3 (4) | 1 (1)
Teething (Gastrointestinal disorders) | 12 (32) | 7 (12) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 48 (91) | 24 (42) | 3 (4) | 6 (6) | 2 (4)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 36 (66) | 23 (35) | 1 (2) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 27 (47) | 7 (16) | 2 (2) | 5 (9) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 10 (17) | 3 (7) | 3 (4) | 2 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 22 (35) | 9 (30) | 3 (7) | 4 (7) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 9 (14) | 2 (3) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 85 (244) | 44 (96) | 4 (14) | 4 (7) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 59 (125) | 30 (67) | 7 (22) | 6 (24) | 2 (4)
Erythema (Skin and subcutaneous tissue disorders) | 36 (49) | 15 (27) | 2 (4) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 37 (55) | 14 (24) | 2 (2) | 4 (17) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (39) | 13 (13) | 3 (4) | 1 (1) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 9 (15) | 6 (7) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 103 (240) | 43 (129) | 13 (27) | 7 (20) | 2 (2)
Nasopharyngitis (Infections and infestations) | 53 (102) | 18 (35) | 2 (11) | 3 (12) | 0 (0)
Viral Infection (Infections and infestations) | 47 (76) | 19 (25) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 31 (41) | 13 (17) | 3 (4) | 1 (1) | 1 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 30 (46) | 13 (21) | 5 (7) | 2 (3) | 1 (2)
Ear Infection (Infections and infestations) | 23 (42) | 15 (28) | 1 (1) | 1 (1) | 2 (3)
Respiratory Tract Infection Viral (Infections and infestations) | 29 (54) | 8 (21) | 2 (5) | 2 (3) | 1 (2)
Gastroenteritis Viral (Infections and infestations) | 23 (24) | 3 (7) | 0 (0) | 0 (0) | 1 (2)
Otitis Media (Infections and infestations) | 21 (33) | 4 (8) | 3 (3) | 3 (3) | 1 (1)
Croup Infectious (Infections and infestations) | 12 (13) | 12 (15) | 0 (0) | 2 (3) | 1 (2)
Influenza (Infections and infestations) | 14 (14) | 5 (6) | 2 (2) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 10 (11) | 7 (12) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 14 (15) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 6 (7) | 2 (2) | 2 (2) | 0 (0)
Otitis Media Acute (Infections and infestations) | 1 (1) | 6 (7) | 1 (1) | 0 (0) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 10 (12) | 12 (18) | 1 (1) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 11 (16) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Eye Swelling (Eye disorders) | 12 (16) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Application Site Rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Application Site Hemorrage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Application Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Application Site Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Application Site Dryness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Irritability Postvaccinal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bullous Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Coxsackie Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail Bed Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perianal Streptococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Circumoral Oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Idiopathic Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis Generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Rash Generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Oral Pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chapped Lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip Pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Allergy To Arthropod Sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atopy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mite Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycotic Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Extra Dose Administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema of Eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood Altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood Swing (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Growth Hormone Deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03211247/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03211247/SAP_001.pdf